CLINICAL TRIAL: NCT05535517
Title: Development and Validation of an Investigator Global Assessment Score for Keratosis Pilaris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Premier Specialists, Australia (Other)
Responsible Party: Principal Investigator, Dedee Murrell, Professor, Director of Premier Specialists, Premier Specialists, Australia
Other Study IDs: KPIGA2022
Record Dates: First submitted 2022-08-30; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Keratosis Pilaris
Keywords: scoring system; IGA score; severity; disease assessment; KP; evaluation
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: KP Scoring Day Participants
  Participants who attend the one-day scoring session in August 2022.
  Interventions: Other: KPAI; Other: KP-IGA
- Group 2: KP Follow-up Scoring (September)
  Participants who attended the scoring day in August will be invited to attend a follow-up scoring session in September - October 2022. The purpose of this scoring session is to see how stable their condition is and take baseline photographs of their skin to monitor their condition.
  Four assessors will score the participants in 5-minute intervals with the proposed scoring system KPAI and the KP-IGA. Participants will be offered free samples of Cerave Salicylic Acid Smoothing Cleanser and Cream to try.
  Interventions: Other: CeraVe SA Smoothing Cleanser; Other: CeraVe SA Smoothing Cream; Other: KPAI; Other: KP-IGA
- Group 3: KP Follow-up Scoring (November)
  Participants who attend the September scoring session will be invited to return for another rescoring in November - December 2022 to see if there is any improvement in their KP and if the score is responsive to change.
  Participants will be given free samples of Propaira 30% Urea exfoliating emollient and Propaira 20% Lactic acid exfoliating lotion to try.
  Interventions: Other: Propaira 20% Lactic Acid Exfoliating Lotion; Other: Propaira 30% Urea Exfoliating Emollient; Other: KPAI; Other: KP-IGA
- Group 4: KP Follow-up Scoring (December)
  Participants who attend the November scoring session will be invited to return for another rescoring in December 2022 to monitor their progress, and see if there is any improvement in their KP and if the score is responsive to change.
  Interventions: Other: KPAI; Other: KP-IGA

INTERVENTIONS:
Other: CeraVe SA Smoothing Cleanser — The CeraVe Salicylic Acid (SA) Smoothing Cleanser is formulated with salicylic acid to help exfoliate the skin and remove dirt and dead skin cells on the skin without compromising or striping moisture from the skin's natural barrier, leaving the skin feeling clean, smooth and hydrated. This salicylic acid cleanser is also formulated to include hyaluronic acid to hydrate and retain moisture and 3 essential ceramides to moisturise and help support the skin's barrier.
  Groups: Group 2
Other: CeraVe SA Smoothing Cream — The CeraVe Salicylic Acid (SA) Smoothing Cream contains salicylic acid as well as hydrating hyaluronic acid and three essential ceramides.
  Groups: Group 2
Other: Propaira 20% Lactic Acid Exfoliating Lotion — For smoothing rough skin.
  Groups: Group 3
Other: Propaira 30% Urea Exfoliating Emollient — 30% Urea, 7% Glycerin to smoothen rough skin.
  Groups: Group 3
Other: KPAI — The proposed score, Keratosis Pilaris Area Index (KPAI), is a 5-point IGA score (0-4) of five main body areas: face, upper limbs, lower limbs, trunk, and buttocks, for a maximum of 20 in two main categories, activity (erythema, skin roughness and papulation) and damage (pigmentation and scarring). The final score will be a maximum of 100.
  Other Names: Keratosis Pilaris Area Index
Other: KP-IGA — A standard 5-point IGA score (0-4) defined specifically for KP

SUMMARY:
This validation study aims to develop a standardised investigator global assessment (IGA) score for keratosis pilaris and test the validity and reliability of the score through a one-day scoring exercise held at a private practice and compare it to a standard 0-4 IGA score specifically defined for keratosis pilaris.

DETAILED DESCRIPTION:
This is a prospective validation study aiming to develop and validate a standardised IGA score for KP. Firstly, a preliminary score will be developed using deidentified photos of patients with KP. These photos will only be used to create the training slide for the assessors. The proposed score, Keratosis Pilaris Area Index (KPAI), is a 5-point IGA score (0-4) of five main body areas: face, upper limbs, lower limbs, trunk, and buttocks, for a maximum of 20 in two main categories, activity (erythema, skin roughness and papulation) and damage (pigmentation and scarring). The final score will be a maximum of 100. This will be compared to a standard 0-4 IGA score, defined specifically for KP, known as a KP-IGA.

The one-day scoring exercise has been modified from the Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) validation (Loh et al., 2014). It will take place at Premier Specialists, Kogarah, Sydney with all co-investigators conducting the study in person at this single study site. Each dermatologist and medical professional involved will receive training on using the scores through a slideshow of training photos prior to the live scoring session. Five dermatologists and four medical professionals will be randomly assigned to assess 20 KP patients in 5-minute intervals, using the proposed scoring system, KPAI, and the KP-IGA score. This data will be used to assess inter-rater reliability.

Each dermatologist or medical professional will be randomly assigned to rescore two patients after seeing other patients to minimise recall bias. The randomisation will be done by an investigator who is uninvolved in the scoring session and has had no interaction with both patients and assessors. Data gathered from this section is used to determine intra-rater reliability.

Every participant will also complete two QOL questionnaires: the DLQI/CDLQI and HADS. This data will be used to provide insight of patient's subjective perceptions of KP and the psychological impact it may have on them.

Participants who attended the scoring day will be invited to attend a follow-up scoring session in September - October 2022. The purpose of this scoring session is to see how stable their condition is and take baseline photographs of their skin to monitor their condition.

Four assessors will score the participants in 5-minute intervals with the proposed scoring system KPAI and the KP-IGA. Participants will be offered free samples of Cerave Salicylic Acid Smoothing Cleanser and Cream to try. They will be invited to return for another rescoring in November - December 2022 to see if there is any improvement in their KP and if the score is responsive to change.

In the November - December 2022 scoring session, participants will be given free samples of Propaira 30% Urea exfoliating emollient and Propaira 20% Lactic acid exfoliating lotion to try. They will be invited to return for a fourth scoring session in December to monitor their progress and see if the scores improve.

ELIGIBILITY:
Inclusion Criteria:

* All genders are allowed to participate
* Age range: 12-80 years
* Those with KP including subtypes of KP
* Able to attend the one-day scoring session
* Participants having read and understood the patient information and consent form and are willing to participate
* Of mature mind and able to provide informed consent, in case of children (< 18 years) then the guardian or caretaker can provide consent
* Able to maintain compliance with required study related procedures including completing the QOL questionnaire's

Exclusion Criteria:

* Participants who are unwilling or unable to attend the one-day scoring session
* Those with other skin conditions overlapping the same area(s) as the KP

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the Principal Investigator's dermatology practice who have been diagnosed with keratosis pilaris.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-08-13 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Keratosis Pilaris Area Index (KPAI) | through study completion, an average of 1 year
  This study aims to develop and validate an IGA score for evaluating KP (KPAI) by determining the intra-rater and inter-rater reliability through testing the composite IGA score on patients and comparing it to a standard 0-4 IGA that will be defined specifically for KP.

SECONDARY OUTCOMES:
QOL questionnaires (DLQI/CDLQI) | through study completion, an average of 1 year
  The secondary aim of the study is to explore the impact KP may have on patients' QOL by using the (Child) Dermatology Life Quality (DLQI/CDLQI) Index questionnaires.
QOL questionnaires (HADS) | through study completion, an average of 1 year
  The secondary aim of the study is to explore the impact KP may have on patients' QOL by using the hospital anxiety and depression scale (HADS) questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Dédée Murrell, Principal Investigator — Premier Specialists
Locations (1):
- Premier Specialists, Kogarah, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loh CC, Kim J, Su JC, Daniel BS, Venugopal SS, Rhodes LM, Intong LR, Law MG, Murrell DF. Development, reliability, and validity of a novel Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI). J Am Acad Dermatol. 2014 Jan;70(1):89-97.e1-13. doi: 10.1016/j.jaad.2013.09.041. PMID 24355263